CLINICAL TRIAL: NCT07271914
Title: Pelvic peritOnectomy iN Early Stage Ovarian Tumors: a prospEctive Study
Brief Title: PONDER: Pelvic Peritonectomy in Early Stage Ovarian Tumors
Acronym: PONDER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Responsible Party: Principal Investigator, Elena Olearo, MD, Ospedale Santa Croce-Carle Cuneo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CnGin20251
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Early Stage Ovarian Tumors; Peritoneal Carcinosis
Keywords: ovarian cancer; early stage; ovarian tumor; peritoneal carcinosis; pathology assessment
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention Model: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled patients with FIGO 2018 IA-IB epithelial or non-epithelial ovarian/fallopian tube neoplasma (Other): All patients will receive standard pre-, intra-, and postoperative care according to institutional guidelines. The peritonectomy procedure will not alter the choice of surgical access. Pelvic peritonectomy specimens will be analyzed as part of the final pathology report.
  Interventions: Procedure: systematic surgical approach to wider peritoneal biopsies according with dissection of retroperitoneal spaces, nerve-sparing approach; Diagnostic Test: Histopathologic Analysis

INTERVENTIONS:
Procedure: systematic surgical approach to wider peritoneal biopsies according with dissection of retroperitoneal spaces, nerve-sparing approach — Surgical Procedure:
  Initial step: Exclude upper abdominal disease through inspection and guideline-based biopsies.
  Pelvic peritoneal resection: En bloc or segmental removal of predefined pelvic peritoneal regions according to dissection of retroperitoneal spaces with a nerve-sparing technique.
Diagnostic Test: Histopathologic Analysis — Fixation: 10% neutral-buffered formalin for 6-48 hours. Processing: Paraffin eembedding and complete sampling for histology. Staining: H&E and immunohistochemistry (MOC-31, BER-EP4) to identify epithelial tumor cells. Reporting: Checklist for peritoneal disease

SUMMARY:
Early-stage ovarian tumors represent approximately 30% of all newly diagnosed ovarian cancers. Current international guidelines recommend random peritoneal biopsies for surgical staging, but the diagnostic yield of these biopsies remains limited. The PONDER study aims to evaluate whether standardized surgical procedure and pathology assessment of wider peritoneal pelvic biopsies can increase the detection rate of microscopic peritoneal implants and micrometastases in patients with early-stage ovarian tumors. This multicenter, prospective, single-arm study includes both minimally invasive and open surgical approaches, with a standardized gross and microscopic evaluation of the resected peritoneal specimens

DETAILED DESCRIPTION:
The study focuses on the excision of anatomically defined pelvic peritoneal areas, with meticulous dissection of the retroperitoneal spaces and a nerve-sparing approach. Combined with a specific pathology protocol, this strategy improves the detection of microscopic peritoneal involvement and provides new insights into the mechanisms of pelvic recurrence

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* FIGO 2018 stage IA-IB epithelial or non-epithelial ovarian or fallopian tube tumors
* Complete preoperative work-up (ultrasound, CT scan, tumor markers)
* Laparoscopic, robotic or open surgical approach
* Signed informed consent

Exclusion Criteria:

* Sarcomas, melanomas, mesotheliomas, hematologic malignancies
* Advanced ovarian tumors
* Fertility-sparing surgery with uterine preservation
* Inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 390 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of positive peritoneal biopsies after pelvic peritonectomy (detection of microscopic implants). | from surgery up to at least 24 months of follow up after surgery
  Proportion of positive peritoneal biopsies after pelvic peritonectomy (detection of microscopic implants)

SECONDARY OUTCOMES:
Perioperative complications | from the date of surgery up to six months after surgery
  Clavien-Dindo classification
Recurrence site | from the date of surgery up to at least 24 months of follow up
2-year progression free survival | 24 months after surgery
2-year overall survival | 24 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Puppo, MD, Principal Investigator — Azienda Ospedaliera Santa Croce e Carle Cuneo; Elena Olearo, MD, Study Director — Azienda Ospedaliera Santa Croce e Carle Cuneo
Locations (1):
- Azienda Ospedaliera Santa Croce e Carle Cuneo, Cuneo, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared with investigators from other centers and results published according to national and international regulatory requirements
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] van de Vorst REWM, Hoogendam JP, van der Aa MA, Witteveen PO, Zweemer RP, Gerestein CG. The attributive value of comprehensive surgical staging in clinically early-stage epithelial ovarian carcinoma: A systematic review and meta-analysis. Gynecol Oncol. 2021 Jun;161(3):876-883. doi: 10.1016/j.ygyno.2021.04.007. Epub 2021 Apr 10. PMID 33849726